CLINICAL TRIAL: NCT07168018
Title: A Phase II Randomised, Open-label Study of the Safety and Immunogenicity of Coadministration of the Candidate Rabies Vaccine ChAdOx2 RabG and Licensed Vaccine
Brief Title: Safety and Immunogenicity of Coadministration of the Candidate Rabies Vaccine ChAdOx2 RabG and Licensed Vaccine
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAB003
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Rabies
Keywords: Vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A1 (Adults) (Experimental): Participants aged 18-45 years will receive coadministration of 5×10^10 vp ChAdOx2 RabG (2 site IM) and licensed IRV (2 site IM) at a single visit. Rabies virus neutralisation antibody (VNA) titres will be determined at baseline and days 7, 14, 21, 28, and 56. Participants will receive a 1-site IM vaccination with IRV on day 56.
  Interventions: Biological: Coadministration of ChAdOx2 RabG and licensed inactivated rabies vaccine (IRV)
- Group A2 (Adults) (Active Comparator): Participants aged 18-45 years will receive a licensed IRV (2 site ID) at days 0, 3 and 7. Rabies virus neutralisation antibody (VNA) titres will be determined at baseline and days 7, 14, 21, 28, and 56.
  Interventions: Biological: Inactivated Rabies Vaccine (IRV)

INTERVENTIONS:
Biological: Coadministration of ChAdOx2 RabG and licensed inactivated rabies vaccine (IRV) — A single visit of coadministration of 5×10^10 vp ChAdOx2 RabG (2 site IM) and licensed IRV (2 site IM).
  Arms: Group A1 (Adults)
Biological: Inactivated Rabies Vaccine (IRV) — A World Health Organization (WHO) prequalified IRV at two anatomical sites (2 site ID) on days 0, 3 and 7.
  Other Names: Verorab
  Arms: Group A2 (Adults)

SUMMARY:
This is a phase II randomised, open-label study to assess the safety and immunogenicity of coadministration of the candidate rabies vaccine ChAdOx2 RabG and licensed vaccine in healthy adults (18-45 years old). ChAdOx2 RabG will be administered intramuscularly and licensed rabies vaccine will be given either intramuscularly (i.e., for the intervention group) or by intradermal injection (i.e., for the control group).

DETAILED DESCRIPTION:
A total of 40 participants will be recruited into 2 groups in Bagamoyo, Tanzania. The duration of the study will be up to 56 days per participant from the time of first vaccination. Participants in the intervention group will receive coadministration of ChAdOx2 RabG and licensed inactivated rabies vaccine (IRV) at a single visit, while participants in the control group will receive only licenced rabies vaccine at 3 visits.

Participant groups who will receive coadministration of ChAdOx2 RabG and licensed rabies vaccine will also receive a 1-site IM vaccination with IRV on day 56.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults aged 18-45 years at the time of enrolment with signed consent.
* (Female only participants): Must be non-pregnant (as demonstrated by a negative serum pregnancy test) and willing to use an effective form of contraception.

  *Female volunteers are required to use an effective form of contraception during the course of the study. There is currently no information about the effect of this vaccine on a foetus. Acceptable forms of contraception for female volunteers include:
* Established use of injected or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Total abdominal hysterectomy.
* Planned long-term (at least 2 months from the date of the first vaccination) or permanent residence in Bagamoyo town.
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2
* Correctly answer all 10 questions on the protocol and study procedures understanding questionnaire within 2 attempts.

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
* Clinically significant history of skin disorder, allergy, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease and neurological illness which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data as judged by the PI or other delegated individual.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including IRVs e.g. amphotericin B, chlortetracycline, neomycin, polymyxin, streptomycin
* Any history of anaphylaxis in relation to vaccination.
* Clinically significant laboratory abnormality as judged by the PI or other delegated individual.
* Receipt of any previous rabies vaccinations, including an incomplete course of IRV and/or any doses of ChAdOx2 RabG.
* History of vaccination with previous adenoviral vectored vaccines in the 6 months prior to enrolment in the study, or of vaccination with any other vaccine (including non-adenovirus-vectored COVID-19 vaccines) in the 28 days prior to enrolment.
* Planned / likely receipt of any other vaccine within 28 days after enrolment.
* History of bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture, or continuous anticoagulation e.g., with warfarin
* History of confirmed major thrombotic event, (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism) or,
* History of antiphospholipid syndrome.
* History of prior receipt of unfractionated heparin
* History of heparin induced thrombocytopenia
* Receipt of any blood products/ immunoglobulins within the three months preceding the planned administration of the vaccine candidate.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG).
* Likelihood of travel away from the study area.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Contraindication to use of paracetamol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of coadministration of ChAdOx2 RabG and inactivated rabies vaccine (IRV) in healthy adults (18-45 years) residing in a rabies endemic country by the occurrence of solicited adverse events. | Assessment of solicited AEs in the first 7 days post vaccination
  Occurrence of local and systemic solicited AEs
Safety and tolerability of coadministration of ChAdOx2 RabG and inactivated rabies vaccine (IRV) in healthy adults (18-45 years) residing in a rabies endemic country by the occurrence of unsolicited adverse events. | Unsolicited AEs to be assessed up to 28 days post vaccination
  Occurrence of unsolicited local and systemic adverse events
Safety and tolerability of coadministration of ChAdOx2 RabG and inactivated rabies vaccine (IRV) in healthy adults (18-45 years) residing in a rabies endemic country by the occurrence of laboratory adverse events. | Clinical laboratory AEs to be assessed up to 28 days post vaccination.
  Occurrence of laboratory adverse events.
Safety and tolerability of coadministration of ChAdOx2 RabG and inactivated rabies vaccine (IRV) in healthy adults (18-45 years) residing in a rabies endemic country by the occurrence of serious adverse events. | SAEs will be collected from enrolment until the end of the follow-up period (Day 56).
  Occurrence of serious adverse events

SECONDARY OUTCOMES:
A comparison of the immunogenicity of a singe-visit IM coadministration of ChAdOx2 RabG and licensed IRV versus three-visit ID administration of licensed IRV. | Rabies virus neutralisation antibody titres will be determined at baseline and days 7, 14, 21, 28, and 56.
  Rabies virus neutralising antibody (VNA) will be assessed by rapid fluorescent focus inhibition test (RFFIT).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Douglas, Principal Investigator — Jenner Institute, University of Oxford
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania